CLINICAL TRIAL: NCT01055301
Title: S0833, Modified Total Therapy 3 (TT3) for Newly Diagnosed Patients With Multiple Myeloma (MM): A Phase II SWOG Trial for Patients Aged ≤ 65 Years
Brief Title: S0833, Bortezomib, Thalidomide, Lenalidomide, Combination Chemotherapy, and Autologous Stem Cell Transplant in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0833; S0833 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma; Plasma Cell Myeloma
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cisplatin; Cyclophosphamide; Dexamethasone; Doxorubicin; Etoposide; Lenalidomide; Melphalan; Thalidomide; Gene Expression Profiling; Microarray Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): Ind (1cycle):
  bort 1mg/m2 IV/SQ D1,4,8,11 D1-4: thalid 200mg/d & dex 20mg/d PO; cisplatin & dox 10mg/m2/d, cyclophos 400mg/m2/d, etoposide 40mg/m2/d contIV; enoxaparin 40mg/d SQ prn.
  PBSC Coll: at recovery per local standard
  Bridging (before/between trans/after Cons):
  thal 50mg/d D1-21 & dex 20mg D1,8,15 PO
  Tandem Trans (x2):
  bort 1mg/m2 IV/SQ D-4,-1 D-4to-1: mel 50 mg/m2 IV, thal 200mg/d & dex 40mg/d PO PBSC >/=200x10^6 cells
  Cons (1cycle):
  same as Ind except cis/dox 7.5mg/m2/d, cyclo 300mg/m2/d, no enox
  Maint(</= 3 yrs):
  D1,8,15,22:bort 1mg/m2 IV/SQ, dex 20mg/d PO; len 20mg/d PO D1-20
  Interventions: Drug: bortezomib; Drug: cisplatin; Drug: cyclophosphamide; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: lenalidomide; Drug: melphalan; Drug: thalidomide; Genetic: gene expression analysis; Genetic: microarray analysis; Other: laboratory biomarker analysis; Procedure: autologous-autologous tandem hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: bortezomib
  Other Names: bort
Drug: cisplatin
Drug: cyclophosphamide
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: lenalidomide
Drug: melphalan
Drug: thalidomide
Genetic: gene expression analysis
Genetic: microarray analysis
Other: laboratory biomarker analysis
Procedure: autologous-autologous tandem hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as thalidomide and lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, cisplatin, doxorubicin hydrochloride, cyclophosphamide, etoposide, and melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Combining chemotherapy with autologous stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Giving bortezomib, thalidomide, and combination chemotherapy before and after transplant and lenalidomide after transplant may be an effective treatment for multiple myeloma.

PURPOSE: This phase II trial is studying how well giving bortezomib, thalidomide, and lenalidomide together with combination chemotherapy and autologous stem cell transplant works in treating patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess progression-free survival (PFS) at 3 years in patients with newly diagnosed multiple myeloma (MM) treated with modified Total Therapy 3 (TT3).

Secondary

* To estimate the frequency and severity of toxicities associated with this treatment strategy in these patients.

Correlative

* To perform gene expression profiling on CD138+ purified MM cells and unseparated bone marrow biopsy samples to identify the bone marrow micro-environment signature.
* To determine whether the 70-gene model, developed in the Arkansas Total Therapy 2 (TT2) and validated in the Arkansas TT3 study, also applies to the cooperative group setting.
* Determine whether the novel finding in TT3 of the prognostically favorable suppression of a micro-environment-associated gene, MAG1, also applies to the cooperative group setting.
* Once in complete remission, determine whether the MAG signatures can return to a normal individual's signature as an indication of profound tumor cytoreduction with durable PFS.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive bortezomib IV on days 1, 4, 8, and 11; oral thalidomide and oral dexamethasone on days 1-4; and cisplatin IV continuously, doxorubicin hydrochloride IV continuously, cyclophosphamide IV continuously, and etoposide IV continuously on days 1-4.
* Peripheral blood stem cell (PBSC) collection: Beginning within 2 months after completion of induction therapy, patients undergo PBSC collection until an adequate number of cells are collected. Patients with persistent disease after completion of induction therapy proceed to bridging therapy after adequate stem cells are collected. Patients not requiring bridging therapy proceed directly to transplant.
* Bridging therapy: Patients receive oral thalidomide on days 1-21 and oral dexamethasone on days 1, 8, and 15. Treatment repeats every 21 days for 1-2 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to transplant.
* First autologous PBSC transplantation: Beginning within 6 weeks to 3 months after completion of induction therapy (or ≥ 1 week after completion of bridging therapy), patients receive bortezomib IV on days -4 and -1 and melphalan IV, oral thalidomide, and oral dexamethasone on days -4 to -1. Patients undergo autologous PBSC transplantation on day 0.
* Inter-transplant bridging therapy: Patients with persistent disease after completion of the first autologous PBSC transplant receive bridging therapy as above and then proceed to the second transplant. Patients not requiring bridging therapy proceed directly to the second transplant.
* Second autologous PBSC transplantation: Beginning within 6 months after the first PBSC transplant, patients receive bortezomib, melphalan, thalidomide, and dexamethasone and undergo autologous PBSC as in the first transplant. Patients who skip the second transplant (due to medical or insurance reasons or refusal) proceed to consolidation therapy.
* Consolidation therapy: Beginning within 6 months after the last transplant, patients receive bortezomib, thalidomide, dexamethasone, cisplatin, doxorubicin hydrochloride, cyclophosphamide, and etoposide as in induction therapy.
* Post-consolidation bridging therapy: Patients with persistent disease after completion of consolidation therapy receive oral thalidomide on days 1-21 and oral dexamethasone on days 1, 8, and 15. Patients then proceed to maintenance therapy. Patients not requiring bridging therapy proceed directly to maintenance therapy.
* Maintenance therapy: Beginning within 4 months after completion of consolidation therapy or post-consolidation bridging therapy, patients receive bortezomib IV and oral dexamethasone on days 1, 8, 15, and 22 and oral lenalidomide on days 1-20. Courses repeat every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.

Blood and bone marrow samples may be collected at baseline and periodically during study for gene expression profile analysis.

After completion of study therapy, patients are followed up periodically for up to 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed active multiple myeloma (MM)
* Measurable disease

  * Non-secretory disease allowed provided patient has ≥ 20% plasmacytosis or multiple (> 3) focal plasmacytomas on skeletal survey and/or MRI

PATIENT CHARACTERISTICS:

* Zubrod performance status (PS) 0-2 (Zubrod PS 3-4 allowed if based solely on bone pain)
* ANC ≥ 1,500/mm^3*
* Platelet count ≥ 150,000/mm^3*
* Serum creatinine clearance of ≥ 60 mL/min

  * Patients with creatinine clearance of < 60 mL/min receive a lower dose of melphalan
  * No patients receiving or planning to receive dialysis
* Total bilirubin ≤ 1.5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

  * Must be fully aware of the teratogenic potential of thalidomide
  * Must be willing to comply with the FDA-mandated S.T.E.P.S. program
* Ejection fraction > 40% as measured by MUGA scan or two-dimensional ECHO
* No peripheral neuropathy ≥ grade 2 per CTCAE v. 4.0
* No known hypersensitivity to bortezomib, boron, or mannitol
* No uncontrolled diabetes defined as fasting glucose level > 200 mg/dL on at least more than two occasions or more that two serum random blood levels > 300 mg/dL despite adequate treatment

  * Patients with a history of diabetes mellitus requiring treatment should be on a stable regimen and have their blood glucose closely monitored
* No other malignancy within the past 5 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment within the past year NOTE: *Unless myeloma-related marrow infiltration is documented, defined as ≥ 30% marrow cellularity with 50% of the cells being malignant plasma cells.

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior chemotherapy or radiotherapy
* No more than 1 prior course of chemotherapy for MM

  * Prior chemotherapy must not have included melphalan
* No prior radiotherapy to large area of the pelvis (more than half of the pelvis)
* Prior radiotherapy for symptomatic localized bone lesions or impending cord compression allowed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 3 years | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Frequency and severity of toxicities | 3 years
Gene expression profiling analysis of CD138+ purified plasma cells | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Muneer H. Abidi, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (21):
- United States (21):
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Hematology-Oncology Clinic, Baton Rouge, Louisiana
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington